CLINICAL TRIAL: NCT00539175
Title: Treatment of Painful Diabetic Neuropathy With Photon Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Bay Institute for Research and Education (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Swislocki-1
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Diabetic Neuropathy, Painful; Diabetic Neuralgia; Diabetic Polyneuropathy; Diabetic Mononeuropathy
Keywords: diabetes mellitus; neuropathy; diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): active treatment with infrared light
  Interventions: Device: infrared light
- 1 (Placebo Comparator): sham (placebo) treatment without infrared light
  Interventions: Device: infrared light; placebo

INTERVENTIONS:
Device: infrared light — pulsed infrared light will be applied to feet, ankles and popliteal fossae of patients with diabetic neuropathy
  Arms: 2
Device: infrared light; placebo — patients will be exposed to the same machine used to provide pulsed infrared light, but the light emitting diodes will not be activated. All other aspects of the treatment will be the same. The patient and investigator will be blind to treatment assignment.
  Arms: 1

SUMMARY:
1. Objectives:

1. To assess the efficacy of Photon Stimulation compared with placebo, in treating the pain of diabetic neuropathy.
2. To show that Photonic Stimulation for the treatment of painful diabetic neuropathy is cost effective compared to traditional medical interventions. The latter will be explored by an extensive search of the literature and from an equal number of patients being treated in traditional medical practices using traditional medical interventions. At the conclusion of the study the data will be analyzed for cost-benefits and the possibility of crafting a best-practices approach to treat these syndromes that cost billions of dollars a year in health care expenses and lost productivity.

2. Research Design

This is a double blinded, randomized, placebo-controlled study of 120 patients with painful diabetic neuropathy. These 120 will be randomly assigned treatments utilizing Photon Therapy, using a defined treatment protocol. We expect that some patients will drop out, and our goal is 100 treated patients, for statistical purposes. The Photon Therapy group will be split into two groups, one group that receives Active Photon Therapy and one group that will be treated with the same type of equipment that has been modified to emit no infrared photons (Non Active Photon Therapy Group ("Placebo")). The patients in the "Non Active Photon Therapy Group" will be offered an Active Photon Treatment Session after completion of the study. The patients in the Photon Therapy Groups will be randomized. There will also be an Historical Control Group of patients, fifty, will have received traditional medical interventions (e.g., narcotics, seizure medications) in traditional medical practices. Data from these individuals will be used to calculate potential cost savings.

3. Methodology:

Subjects who meet the inclusion and exclusion criteria and have signed a valid informed consent will be eligible to participate in the study. After screening, subjects in the Photon Therapy groups (both active and nonactive) will undergo four treatment sessions. The first treatment session will vary from the second, third and fourth. During all treatment session, each patient will be imaged with the TIP Infrared Camera before, and after treatment. Infrared imaging can visualize skin temperature changes in a noninvasive manner (2). The first treatment will utilize slightly different protocol than subsequent visits, reduced Photon dosage, 120 instead of 240 joules. Proprioception and protective sensation, characterized by the Semmes-Weinstein monofilament test, and visual and analog pain scoring will also be evaluated before and after each Photon Therapy treatment.

4. Finding:

To date, we have just completed 120 patients, using a block randomization scheme not previously reported in this field. We have collected data on nerve function, pain, quality of life, and skin circulation. The data will remain stored until the study is complete to preserve the blinded nature of the project. Data analysis is still incomplete.

4. Clinical Significance

Diabetic neuropathy is a chronic and progressive condition that potentially leads to disabling pain, and worse, amputation, for many individuals in the United States each year. Present treatments utilize antiseizure medications, opiate analgesics, and antidepressants, and are inconsistently effective. Development of a new treatment strategy potentially could have significant benefit for a great many patients.

DETAILED DESCRIPTION:
• PURPOSE, METHODS, AND PROCEDURES:

1. Purpose:

1. To assess the efficacy of Photon Stimulation compared with placebo, in treating the pain of diabetic neuropathy.
2. To show that Photonic Stimulation for the treatment of painful diabetic neuropathy is cost effective compared to traditional medical interventions. The latter will be explored by an extensive search of the literature and from an equal number of patients being treated in traditional medical practices using traditional medical interventions. At the conclusion of the study the data will be analyzed for cost-benefits and the possibility of crafting a best-practices approach to treat these syndromes that cost billions of dollars a year in health care expenses and lost productivity.

2. Methods

This is a double blinded, randomized, placebo-controlled study of approximately 170 patients with painful diabetic neuropathy. The study sample size is 170 patients. Of these 120 will be given treatments utilizing Photon Therapy, using a defined treatment protocol. We plan to recruit 120 patients to allow for drop out, and to provide 100 completed patients, as requested by FDA. The Photon Therapy group will be split into two groups, one group that receives Active Photon Therapy and one group that will be treated with the same type of equipment that has been modified to emit no infrared photons (Non Active Photon Therapy Group ("Placebo")). The patients in the "Non Active Photon Therapy Group" will be offered an Active Photon Treatment Session after completion of the study. The patients in the Photon Therapy Groups will be randomized. The Historical Control Group of patients, fifty, will have received traditional medical interventions (e.g., narcotics, seizure medications) in traditional medical practices.

3. Procedures: Subjects who meet the inclusion and exclusion criteria and have signed a valid informed consent will be eligible to participate in the study. After screening, subjects in the Photon Therapy groups (both active and nonactive) will undergo four treatment sessions. The first treatment session will vary from the second, third and fourth. During all treatment session, each patient will be imaged with the TIP Infrared Camera before, and after treatment. Infrared imaging can visualize skin temperature changes in a noninvasive manner (2). The first treatment will utilize slightly different protocol than subsequent visits, reduced Photon dosage, 120 instead of 240 joules. Proprioception and protective sensation, characterized by the Semmes-Weinstein monofilament test, and visual and analog pain scoring will also be evaluated before and after each Photon Therapy treatment.

* SUBJECT SELECTION: Subjects were initially recruited from the PI's clinic, from a list of patients diagnosed by Dr. Beckley (Electromyographer) with painful diabetic neuropathy, and from local referrals. In October 2004, we received permission to post flyers and solicit patients (identified by Dr Beckley) from primary providers (flyer and letter attached). We also recruited by posting flyers in VANCHCS facilities, and with VANCHCS diabetes educators. Word of mouth also provided many subjects. In September 2006 we modified the flyer to reflect a focused recruitment at Mather. Vulnerable populations will not be studied.
* RISKS: The potential risks to subjects include physical, psychological, social and economic. These are not likely: The physical risks include discomfort from the photon machine. The psychological risks include boredom. The social risks include being labeled as having a chronic illness, and the risk of loss of privacy. The economic risk includes time off from work that may be needed to participate in the treatment program. Confidentiality will be maintained as much as possible, by storing paper data in locked offices, without name identifiers, and electronic data on spreadsheets on password-protected computers in locked offices.
* BENEFITS: Individual subjects may derive benefit via pain relief; this would also obtain to the whole group of patients with painful diabetic neuropathy.
* RISK-BENEFIT RATIO: The risk is minimal, and the benefit minimal to moderate (potentially greater).
* SAFETY MONITORING: Research staff will monitor for safety.
* INFORMED CONSENT PROCEDURES: The PI (Dr. Swislocki) and his staff (Ms. Orth, Ms. Weisshaupt) will conduct, obtain, and document informed consent within VANCHCS facilities.
* PRIVACY AND CONFIDENTIALITY PROTECTIONS: Confidentiality will be maintained as much as possible, by storing paper data in locked offices, without name identifiers, and electronic data on spreadsheets on password-protected computers in locked offices.
* COSTS TO SUBJECTS: No added expenses are expected. No compensation is proposed.
* DISCLOSURE OF PERSONAL AND FINANCIAL INTEREST IN THE RESEARCH STUDY AND SPONSOR: The Principal Investigator has no personal or financial interests in the research or personal or financial interest in the entity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus with painful neuropathy, defined as foot pain >/ 3 on a 0-10 numeric rating scale, chronic foot pain of at least 6 months' duration, and pain characterized as burning, shooting, or stabbing in nature.
* Patients needed to have capacity to provide informed consent and be able to make serial visits for scheduled treatments.

Exclusion Criteria:

* A history of peripheral vascular disease
* Vitamin B12 deficiency
* Low back pain with radiculopathy; Or
* Another painful condition that was difficult to distinguish from painful diabetic peripheral neuropathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-10; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
pain intensity | 1 week

SECONDARY OUTCOMES:
Semmes-Weinstein sensation, proprioception, quality of life | one week

CONTACTS AND LOCATIONS:
Overall Officials: Arthur LM Swislocki, MD, Principal Investigator — VA Northern California Health Care System; UC Davis School of Medicine
Locations (1):
- VA Northern California Health Care System, Martinez, California, United States